CLINICAL TRIAL: NCT03248843
Title: A Phase I, Open Label, Dose Escalation Study of The Safety and Pharmacokinetics of Anti-PD-L1 Monoclonal Antibody KN035 Administered in Subcutaneous Injection as A Single Agent to Japanese Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of PD-L1 Antibody KN035 in Japanese Subjects With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 3D Medicines (Sichuan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: 3D Medicines (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN035-JP-001
Record Dates: First submitted 2017-08-07; First posted 2017-08-14 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: KN035; Solid tumors; Phase 1
MeSH Terms: interventions — envafolimab

STUDY DESIGN:
Intervention Model Description: Cohorts of 3-6 subjects will be enrolled sequentially at escalating doses of 1.0, 2.5, 5.0 and 10 mg/kg of KN035 weekly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KN035 (Experimental): Cohorts of 3-6 subjects will be enrolled sequentially at escalating doses of 1.0, 2.5, 5.0 and 10 mg/kg weekly. Dose escalation will continue until identification of MTD up to a maximum dose of 10 mg/kg.
  Interventions: Drug: KN035

INTERVENTIONS:
Drug: KN035 — Four cohorts dosed at 1.0 mg/kg, 2.5 mg/kg, 5.0 mg/kg, and 10 mg/kg weekly. All cohorts are administered by subcutaneous injection (SC).

SUMMARY:
This is an open label, dose escalation study to evaluate the safety and tolerability of KN035 in Japanese patients with advanced and metastatic solid tumor. The dose escalation will follow the widely used 3+3 design.

DETAILED DESCRIPTION:
This is an open label, dose escalation study to evaluate the safety and tolerability of KN035 in Japanese patients with advanced and metastatic solid tumor.

The dose escalation will follow the widely used 3+3 design. Cohorts of 3-6 subjects will be enrolled sequentially at escalating doses of 1.0, 2.5, 5.0 and 10 mg/kg weekly. Dose escalation will continue until identification of MTD up to a maximum dose of 10 mg/kg. MTD is defined as the highest dose studied at which no more than 1 of 6 subjects has experienced a dose-limiting toxicity (DLT) in Cycle 1. The enrolled patients are managed under hospitalization for DLT observation period (C1 28 days). If no DLTs occur in a cohort of 3 subjects, a new cohort of 3 subjects will be treated at the next higher dose level. If 1 of 3 subjects in a cohort experiences a DLT, that cohort will be expanded to 6 subjects. If only 1 of the 6 subjects has a DLT, then the next cohort of 3 subjects will be treated at the next higher dose level. If 2 or more DLTs occur within a cohort, then that dose level will be above the MTD, and the previous lower (tolerated) dose level will be considered the MTD if ≤ 1 in 6 subjects has a DLT.

A subject who withdraws from the study during Cycle 1 for reasons other than a DLT will be replaced.

Subjects will be monitored for safety and efficacy throughout the study. After radiological tumor assessment at Screening, the first radiological assessment of tumor response status will be performed at Week 12 (± 1 week), unless there is clinical indication warranting earlier radiologic imaging. The same imaging technique used at baseline has to be used throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a histological or cytological diagnosis of any type of carcinoma, progressive metastatic disease, or progressive locally advanced disease not amenable to local therapy. Subjects must have no standard anti-cancer therapy option, who failed established standard medical anti-cancer therapies for a given tumor type.
* Subject is male or female and ≥ 18 years of age on the day of signing informed consent. However, in case a subject is younger than 20 years old, written informed consent will be obtained from both a subject and a legal representative.
* Subject must have a performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Subject must have adequate hematologic and organ function.
* Subject has voluntarily agreed to participate by giving written informed consent.
* Women able to get pregnant has a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the subject to be eligible.
* Female subjects enrolled in the study must be willing to use either 2 adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy or to abstain from heterosexual activity throughout the study, starting with Informed Consent through 120 days after the last dose of study therapy. Women who have had a surgical hysterectomy and/or bilateral oophorectomy, or who are postmenopausal and have not had a menstrual cycle for 12 consecutive months without medical/medicinal reasons are not considered to be of childbearing potential. Approved contraceptive methods include for example; intra uterine device, diaphragm with spermicide*, cervical cap* with spermicide*, male condoms, or female condom *with spermicide* and hormonal method of contraception. Spermicides alone are not an acceptable method of contraception. *: not approved/certified in Japan.

Male subjects must agree to use an adequate method of contraception starting with Informed Consent through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Subject who not recovered from the effects of any prior chemotherapy, radioactive, or biological cancer therapy prior to the first dose of study therapy (for prior cancer therapy drugs, a washout of 5 half-lives or 28 days whichever is shorter is required), or who has not recovered to CTCAE Grade 1 or better from the adverse events due to cancer therapeutics administered more than 4 weeks earlier. Subject who has had erlotinib, gefitinib, afatinib, or crizotinib within 1 week prior to the first dose of study therapy, or who has not recovered to CTCAE Grade 1 or better from the adverse events due to any of these drugs administered more than 1 week earlier. Grade 2 alopecia is allowed to enter.
* Subject is expected to require any other form of antineoplastic therapy while on study (including maintenance therapy with another agent for NSCLC).
* Subject had prior treatment targeting PD-L1. Subjects with prior treatment targeting PD-1 are allowed to enroll if the subject has a washout time of at least 4 weeks. Examples of such anti-PD-L1 agents include (but are not limited to): BMS-936559 (MDX 1105); MPDL3280A (RG7446); and MEDI4736.
* Subject has a medical condition that requires chronic systemic steroid therapy or requires any other form of immunosuppressive medication. However, subjects using physiologic replacement doses of hydrocortisone, or its equivalent, will be considered eligible for this study: up to 20 mg of hydrocortisone (or 5 mg of prednisone) in the morning and 10 mg of hydrocortisone (or 2.5 mg of prednisone) in the evening. Topical, intraocular, and intranasal steroids are allowed.
* Subject has risk factors for bowel obstruction or bowel perforation (examples include but not limited to a history of acute diverticulitis, intra-abdominal abscess, or abdominal carcinomatosis).
* Subject has a known history of a hematologic malignancy, malignant primary brain tumor or malignant sarcoma, or of another malignant primary solid tumor, unless the subject has undergone potentially curative therapy with no evidence of that disease for 5 years.
* Subject has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks prior to study entry, have no evidence of new or enlarging brain metastases and are off steroids for at least 7 days from first dose of KN035.
* Subject previously had a severe hypersensitivity reaction to treatment with another mAb.
* Subject has a history of pneumonitis or interstitial lung disease irrespective of causes (For the purpose of screening of interstitial lung disease, chest X-ray, Sialylated carbohydrate antigen (KL-6) (hereafter, KL-6), percutaneous arterial blood oxygen saturation (hereafter, SpO2) and auscultation are conducted).
* Subject has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism that is stable on hormone replacement will not be excluded from the study.
* Subject has an active infection requiring therapy.
* Subject is positive for Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), active hepatitis B (HBsAg reactive) or hepatitis C (HCV RNA (qualitative) is detected); subjects with negative hepatitis C antibody testing may not need RNA testing.
* Subject has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
* Subject has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Subject has a marked baseline prolongation of QT/QTc (Fridericia's formula) interval (e.g., repeated demonstration of a QTc interval >450 milliseconds (ms) as a guidance considering the patient's background of physiological conditions), or a history of additional risk factors for torsade de pointes (TdP, e.g., heart failure, hypokalemia, family history of Long QT Syndrome), or is using concomitant medications that prolong the QT/QTc interval.
* Subject is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).
* Subjects with symptomatic ascites or pleural effusion. A subject who is clinically stable following treatment for these conditions (including therapeutic thoraco- or paracentesis) is eligible.
* Subject is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study. However, breastfeeding female subject who stopped breastfeeding can be included only if she agrees to stop breastfeeding during the treatment of the investigational drug and to restart breastfeeding 120 days after the last dose of the investigational drug.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities | From screening to up to cycle 1 (28 days)
KN035 safety and tolerability assessed by monitoring AEs per the NCI-CTC-AE Version 4.03, physical examination, electrocardiograms, laboratory measurements and severity of adverse events | From screening to up to 1 months after the last dose of study drug (up to approximately 2 years
  The safety of KN035 will be assessed throughout the study by monitoring adverse events (AEs) per the NCI-CTC-AE Version 4.03, physical examination, electrocardiograms, laboratory measurements and severity of adverse events.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of KN035 in Japanese patients | From Pre-dose of the first dose to up to 48 weeks
Peak Time (Tmax) of KN035 in Japanese patients | From Pre-dose of the first dose to up to 48 weeks
Area under the plasma concentration versus time curve (AUC) of KN035 in Japanese patients | From Pre-dose of the first dose to up to 48 weeks
t1/2 of KN035 in Japanese patients | From Pre-dose of the first dose to up to 48 weeks
Trough concentration of KN035 in Japanese patients | From Pre-dose of the first dose to up to 48 weeks
Plasma clearance (CL) of KN035 in Japanese patients | From Pre-dose of the first dose to up to 48 weeks
Apparent volume of distribution of KN035 in Japanese patients | From Pre-dose of the first dose to up to 48 weeks
Accumulation rate of KN035 in Japanese patients | From Pre-dose of the first dose to up to 48 weeks
Anti-Drug Antibody of KN035 in Japanese patients | From Pre-dose of the first dose to up to 48 weeks
Changes of lymphocyte Subtyping | From Pre-dose of the first dose to up to 48 weeks
Changes of cytokine | From Pre-dose of the first dose to up to 6 months
Objective Response Rate (ORR) | Up to 2 approximately years
Disease Control Rate (DCR) | Up to 2 approximately years
Progression-Free survival (PFS) | Up to 2 approximately years
Duration of Response (DOR) | Up to 2 approximately years

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - St. Marianna University School of Medicine Hospital, Kawasaki
  - National Cancer Center Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cui C, Wang J, Wang C, Xu T, Qin L, Xiao S, Gong J, Song L, Liu D. Model-informed drug development of envafolimab, a subcutaneously injectable PD-L1 antibody, in patients with advanced solid tumors. Oncologist. 2024 Sep 6;29(9):e1189-e1200. doi: 10.1093/oncolo/oyae102. PMID 38982653
- [Derived] Shimizu T, Nakajima TE, Yamamoto N, Yonemori K, Koyama T, Kondo S, Sunakawa Y, Izawa N, Horie Y, Xiang S, Xu S, Qin L, Gong J, Liu D. Phase I study of envafolimab (KN035), a novel subcutaneous single-domain anti-PD-L1 monoclonal antibody, in Japanese patients with advanced solid tumors. Invest New Drugs. 2022 Oct;40(5):1021-1031. doi: 10.1007/s10637-022-01287-7. Epub 2022 Aug 6. PMID 35932387